CLINICAL TRIAL: NCT06894641
Title: A Randomized Control Trial of Enhanced Cognitive Behavioural Group Therapy for Older Adults with Depression: Efficacy Across Older Age-Groups
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Keri-Leigh Cassidy, Professor, Geriatric Psychiatrist, Nova Scotia Health Authority
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 66920
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Major Depression
Keywords: CBT; CBT-OA; Depression; Major Depression; Major Depressive Disorder; Cognitive Behavior Therapy; Older Adults
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Cognitive Behavioral Therapy; Aging

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT-OA Group Therapy (Active Comparator): Participants in this group receive 8 weeks of Cognitive Behavior Therapy for Older Adults (CBT-OA) from study clinicians
  Interventions: Behavioral: Cognitive Behavior Therapy for Older Adults (CBT-OA)
- Treatment As Usual (TAU) (No Intervention): Individual routine care offered by the referring geriatric psychiatrist or the family physician attending to the patient.

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy for Older Adults (CBT-OA) — CBT-OA integrates modifications to standard CBT to consider age-related physical, cognitive and psychological changes. CBT-OA also integrates positive psychiatry principles for older adults to promote behavioural change and health attitude change.
  Arms: CBT-OA Group Therapy

SUMMARY:
This study is on a type of psychotherapy to treat depression in older adults called Cognitive Behavioural Therapy (CBT-OA). CBT is based on the idea that changing thoughts and behaviours can improve mood. CBT has been shown to treat depression in many types of people. CBT-OA changes the usual approaches used for older adults and offers the therapy in a group settings for 8 weeks, for 2 hours a week.

Participants will be randomly (by chance) placed into one of two study groups. One group will receive CBT-OA treatment right away. The other group (Treatment As Usual) will receive standard care from their doctor during the 12-week study period. Both groups will be closely monitored during the study period. The standard care group will be offered CBT-OA in a future session outside of the study.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients 65+ years of age and diagnosed with MDE per DSM-V criteria by a geriatric psychiatrist using a standard clinical biopsychosocial assessment and a Beck Depression Inventory (BDI) of >12.

Exclusion Criteria:

* Patients with psychosis, those undergoing acute inpatient care or electroconvulsive therapy (ECT), those with dementia (Mini-Mental Status Examination (MMSE) score of < 26), and those with chronic personality disorders

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | 12 weeks
  The primary outcome measure will be patient-rated depression on the Beck Depression Inventory-II (BDI-II), a standardized patient-report scale commonly used in CBT depression intervention research.

IPD SHARING:
Plan to Share IPD: No